CLINICAL TRIAL: NCT06136260
Title: The Grief Navigation Trial: A Multi-Site Pragmatic Comparative Effectiveness Trial of Interventions to Support Parents After Their Child's Unexpected or Traumatic Death
Brief Title: The Grief Navigation Trial: A Comparison of Two Interventions to Support Parents After Their Child's Unexpected or Traumatic Death
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Chicago (Other); Patient-Centered Outcomes Research Institute (Other); Missing Pieces, a program of the HAP Foundation (Unknown)
Responsible Party: Principal Investigator, Kelly Michelson, Attending Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-6458
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Bereavement
Keywords: grief; caregivers; community resources; pediatric; self-efficacy; coroners and medical examiners

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization will occur after a medical examiner or coroner (ME) case is referred to Missing Pieces. Participants and MEs will be blinded to participants' treatment arm; Missing Pieces and study staff will be aware of intervention assignments. Missing Pieces will randomize all referred ME cases, (except cases referred from Lake County where the intervention has already been adopted into practice) to CRx-B or GBSI using the method of permuted blocks and the uniform random number function in Stata V17. To ensure balance of intervention arms by ME office, randomization will be stratified by ME office.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CommunityRx-Bereavement (CRx-B) (Experimental)
  Interventions: Other: CommunityRx-Bereavement
- General Bereavement Support Information (GBSI) (Active Comparator)
  Interventions: Other: General Bereavement Support Information

INTERVENTIONS:
Other: CommunityRx-Bereavement — The medical examiner or coroner will refer parents to an organization called Missing Pieces. Missing Pieces does not deliver healthcare services to grieving families; rather, Missing Pieces helps families find grief services in their community.
  For CRx-B, a Grief Navigator from Missing Pieces will text and/or call the parent after receiving the referral; share information about grief and support resources; learn what resources the parent needs for themselves and their family; send the parent a personalized list of grief and social support community resources called a HealtheRx via text, email, or mail; and plan future text message communications with bidirectional functionality and, if requested, subsequent calls or texts from the Grief Navigator to occur at least 3, 6, and 12 months after the child's death.
  Other Names: CRx-B
  Arms: CommunityRx-Bereavement (CRx-B)
Other: General Bereavement Support Information — The medical examiner or coroner will refer parents to an organization called Missing Pieces. Missing Pieces does not deliver healthcare services to grieving families; rather, Missing Pieces helps families find grief services in their community.
  For GBSI, Missing Pieces sends parents a unidirectional text message providing a link to a webpage with a general list of grief resources (e.g., support groups) and information about grief and bereavement within two weeks of the child's death and again 3, 6, and 12 months after the child's death.
  Other Names: GBSI
  Arms: General Bereavement Support Information (GBSI)

SUMMARY:
Parents of children who die traumatically or unexpectedly from things like suicide or an overdose suffer from mental and physical health problems and can experience massive disruptions in their family life. For about half of these parents, the first, and sometimes only, interactions they have with the healthcare system when their child dies are with a medical examiner or coroner (hereafter 'ME'). But MEs have little to no training in helping grieving families, and there are no standards guiding medical examiners or coroners on how or even if they should help grieving families. This gap leaves parents to find the help they need on their own. This research will test two different strategies for addressing this gap in the healthcare system.

DETAILED DESCRIPTION:
Of approximately 60,000 annual deaths of people < 25 years old, ~45% occur unexpectedly or traumatically (e.g., from homicide, suicide, or unintentional injury) and become a medical examiner or coroner (hereafter 'ME') case. Parents and caregivers (hereafter 'parents') of these children suffer debilitating mental health issues like complicated grief and depression, physical problems and family dysfunction, and struggle to find support. Often, the ME is parents' sole point of contact with the healthcare system. Yet MEs have limited education, guidance, and tools to support bereaved parents. Scalable systems-level interventions are needed, at the point of ME care, to connect bereaved parents to critical supports.

This study will compare two interventions to facilitate care across healthcare settings for bereaved parents:

1. CommunityRx-Bereavement (CRx-B), an evidence- and theory-based, low intensity, highly scalable intervention, and
2. General bereavement support information (GBSI), a standardized treatment regimen developed from extant literature and current recommended standards for supporting parents after a child's death.

This is a pragmatic, multi-site 1:1 randomized controlled comparative effectiveness study using a type I hybrid design. CRx-B and GBSI will be carried out by Missing Pieces, a community-based organization. To learn about which strategy works better, the study team will ask parents to complete surveys ~6.5 months after their child dies.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers of ME cases involving a person < 25 years old from one of the following offices: Cook County Medical Examiners, Lake County Coroners, DuPage County Coroner, Will County Coroner, McHenry County Coroner, Kane County Coroner, Peoria County Coroner
* Parents or caregivers who provide permission to the ME to be referred to Missing Pieces
* Parent or caregivers who are referred to Missing Pieces by a ME
* Parents or caregivers able to read and communicate in English or Spanish

Exclusion Criteria:

* Parents or caregivers unable to read or communicate in English or Spanish
* Parents or caregivers under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Parent Self-efficacy for Finding Resources | ~6.5 months after child's death
  Domain-specific item assessing self-efficacy related to support after a child's death, based on Bandura's Self-Efficacy Scale, "How confident are you in your ability to find resources to support you after your child's death?" Responses are on a 5-point Likert scale ranging from "not at all confident" to "completely confident."
Complicated Grief | ~6.5 months after child's death
  Index of Complicated Grief, 19-item tool that uses a 5-point Likert scale ("never" to "always"). Responses are scored 0 to 4 and totaled (0 to 76) with higher scores indicating more symptoms of grief.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Michelson, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Stacy Lindau, MD, MAPP, Principal Investigator — University of Chicago
Locations (7):
- United States (7):
  - Cook County Medical Examiner's Office, Chicago, Illinois
  - Will County Coroner's Office, Joliet, Illinois
  - Peoria County Coroner's Office, Peoria, Illinois
  - Kane County Coroner's Office, Saint Charles, Illinois
  - Lake County Coroner's Office, Waukegan, Illinois
  - DuPage County Coroner's Office, Wheaton, Illinois
  - McHenry County Coroner's Office, Woodstock, Illinois

IPD SHARING:
Plan to Share IPD: Yes
A full data package with the combined data will be created for the purpose of data sharing. During the study period (including data collection and analysis) access to the data will be restricted to the study team. Any secondary analysis of the dataset during the study period will need to be assessed and approved by the dual PIs, Dr. Michelson and Dr. Lindau with input from the steering committee at their discretion. This data package will be uploaded to a HIPAA-compliant, secure file sharing platform hosted by Lurie Children's Hospital and maintained by Lurie Children's Hospital for at least 7 years per PCORI requirements. Lurie Children's Hospital will be responsible for responding to Data Sharing related inquiries.
Time Frame: After the study period for at least 7 years

REFERENCES:
- [Derived] Agha E, Sutter C, Ojewuyi I, Abramsohn EM, Andriano M, Bell C, Calix AL, Cherry JL, Downing K, Flower T, Halm M, Hayes A, Heffernan ME, Hill J, Hoeppner CZ, Jacobson M, Jennings J, Kula-Leitner L, Lee S, Major DR, Makelarski JA, Maruyama NL, McNicholas A, Newton S, Shuber C, Vesco AT, Lindau ST, Michelson KN; Grief Navigation Trial Study Team. The Grief Navigation Trial: A multi-site pragmatic comparative effectiveness trial of two interventions to support parents after their child's unexpected or traumatic death. Contemp Clin Trials. 2025 Aug;155:107962. doi: 10.1016/j.cct.2025.107962. Epub 2025 May 26. PMID 40436312